CLINICAL TRIAL: NCT05909553
Title: A Phase 1, Open-Label Study to Evaluate the Effect of Crushing and Grinding on the Bioavailability of Venetoclax Tablet in Healthy Adult Female Subjects
Brief Title: Study to Assess Adverse Events and Compare How Crushed, Ground, and Intact Oral Tablets Venetoclax Moves Through the Body of Healthy Female Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M24-301
Record Dates: First submitted 2023-06-12; First posted 2023-06-18 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Venetoclax; ABT-199
MeSH Terms: interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Venetoclax Sequence 1 (Experimental): Participants will receive whole venetoclax, followed by crushed venetoclax, and completed with ground venetoclax for a 15 day period.
  Interventions: Drug: Venetoclax
- Venetoclax Sequence 2 (Experimental): Participants will receive crushed venetoclax, followed by ground venetoclax, and completed with whole venetoclax for a 15 day period.
  Interventions: Drug: Venetoclax
- Venetoclax Sequence 3 (Experimental): Participants will receive ground venetoclax, followed by whole venetoclax, and completed with crushed venetoclax for a 15 day period.
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — Oral; Tablet
  Other Names: ABT-199; Venclaxta

SUMMARY:
The objective of this study is to assess the oral bioavailability of crushed and ground venetoclax commercial tablets relative to the intact venetoclax commercial tablets under fed condition in healthy female participants.

ELIGIBILITY:
Inclusion Criteria:

* Must either be: postmenopausal, permanently surgically sterile, or perimenopausal or premenopausal and practicing a method of birth control until at least 1 month after the last dose of study drug.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG).

Exclusion Criteria:

* Significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, cardiovascular, pulmonary or hepatic disease within the past 6 months that in the opinion of the investigator would adversely affect her participating in this study.
* History of any clinically significant sensitivity or allergy to any medication or food.
* History of or active medical condition(s) or surgical procedure(s) that might affect gastrointestinal motility, pH, or absorption.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events | Up to 75 Days
  An adverse event is defined as any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Maximum Observed Plasma Concentration (Cmax) of Venetoclax | Up to 45 Days
  Cmax of venetoclax.
Time to Cmax (Tmax) of Venetoclax | Up to 45 Days
  Tmax of venetoclax.
Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to the Time of the Last Measurable Concentration (AUCt) of Venetoclax | Up to 45 Days
  AUCt of venetoclax.
AUC From Time 0 to the Time Infinity (AUCinf) of Venetoclax | Up to 45 Days
  AUCinf of venetoclax.
Apparent Terminal Phase Elimination Rate Constant (β) of Venetoclax | Up to 45 Days
  Apparent terminal phase elimination rate constant of venetoclax.
Terminal Phase Elimination Half-life (t1/2) of Venetoclax | Up to 45 Days
  T1/2 of venetoclax.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 255783, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alaei S, Wang Y, Liu Y, Schiele J, Deng R, Shiller D, Marroum P, Menon R, Salem AH. Venetoclax Clinical Pharmacokinetics After Administration of Crushed, Ground or Whole Tablets. Clin Ther. 2024 Oct;46(10):752-758. doi: 10.1016/j.clinthera.2024.03.012. Epub 2024 May 22. PMID 38782609
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-301